CLINICAL TRIAL: NCT02276534
Title: SENSE Theatre Research Program
Brief Title: SENSE Theatre Intervention for Children With Autism Spectrum Disorder (ASD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Blythe Corbett, Associate Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 110082
Record Dates: First submitted 2014-10-15; First posted 2014-10-28 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Theatre (Experimental): The participants will receive 10 sessions of peer-mediated, theatre-based intervention.
  Interventions: Behavioral: SENSE Theatre
- No Intervention then Theatre (Experimental): The participants will not receive the treatment for a period of time.
  Interventions: Behavioral: Delayed Intervention

INTERVENTIONS:
Behavioral: SENSE Theatre — A peer-mediated, theatre-based intervention.
  Arms: Theatre
Behavioral: Delayed Intervention
  Arms: No Intervention then Theatre

SUMMARY:
The investigator's goal is to address the need for the development of social interventions for youth with autism in an innovative intervention, SENSE Theatre. The intervention blends established behavioral strategies with theatre techniques that emphasize the involvement of peers, play and performance. The resulting synergy extends promising pilot studies in a randomized group experiment.

DETAILED DESCRIPTION:
The investigator's goal is to address the need for the development of social interventions for youth with autism in an innovative intervention, SENSE Theatre. The intervention blends established behavioral strategies with theatre techniques that emphasize the involvement of peers, play and performance. The resulting synergy extends promising pilot studies in a randomized group experiment.

Objectives: The purpose of the study is to evaluate and extend the impact of a peer-mediated, theatre-based intervention on children with ASD with an emphasis on social functioning. The 10-session program incorporates theatrical approaches, trained typically developing peers and established behavioral strategies. Previous studies using pre-post designs have reported improvement in several skills, such as face memory, theory of mind and social cognition. A primary objective of this investigation is to utilize a true experimental design while evaluating social ability across multiple levels of analysis including neuropsychological, cognitive, behavioral, and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* children diagnosed with autism spectrum disorder with IQ ≥ to 70.

Exclusion Criteria:

* IQ ≤ 70, children with current aggression toward self or others.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2014-08; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
NEPSY Memory for faces | Change from Baseline at Week 10 and Week 16
  The measure requires the child to observe 16 faces of children and then remember them immediately and following a 30-minute delay. Raw scores are generated which are converted to standardized scores based on normative data.
Measurement of Salivary Cortisol levels | Change from Baseline Cortisol level at 20 minutes, 40 minutes, 60 minutes
Event Related Potentials (ERP) incidental memory task | Change from baseline at Week 10 and Week 16
Social Responsiveness Scale | Change from baseline at Week 10 and Week 16
Peer Interaction Playground Paradigm | Change from baseline at Week 10 and Week 16
  A playground play session conducted with trained typically developing peers.
Adaptive Behavior Assessment System | Change from baseline at Week 10 and Week 16
  Parent questionnaire of child's adaptive behavior
Parenting Stress Index | Change from baseline at Week 10 and Week 16
  parent-based questionnaire

SECONDARY OUTCOMES:
Clinical Evaluation of Fundamentals Recalling Sentences subtest | Change from baseline at Week 10 and Week 16
Peabody Picture Vocabulary Test | Change from baseline at Week 10 and Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Blythe A Corbett, Ph.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt Kennedy Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Key AP, Corbett BA. The Unfulfilled Promise of the N170 as a Social Biomarker. Biol Psychiatry Cogn Neurosci Neuroimaging. 2020 Mar;5(3):342-353. doi: 10.1016/j.bpsc.2019.08.011. Epub 2019 Sep 13. PMID 31679960
- [Derived] Corbett BA, Ioannou S, Key AP, Coke C, Muscatello R, Vandekar S, Muse I. Treatment Effects in Social Cognition and Behavior following a Theater-based Intervention for Youth with Autism. Dev Neuropsychol. 2019 Oct;44(7):481-494. doi: 10.1080/87565641.2019.1676244. Epub 2019 Oct 7. PMID 31589087